CLINICAL TRIAL: NCT06901427
Title: Effectiveness of Lifestyle Modification Program on the Quality of Life in Patients with Pemphigus
Brief Title: Impact of a Lifestyle Program on Quality of Life in Pemphigus Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHAbdelhafeez, LECTURER assistant, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Lifestyle in pemphigus
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pemphigus Disease
Keywords: lifestyle, quality of life, pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Diet, Mediterranean; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifestyle Modification Program (Experimental)
  Interventions: Behavioral: Mediterranean Diet and exercise

INTERVENTIONS:
Behavioral: Mediterranean Diet and exercise — A structured dietary intervention promoting Mediterranean-style eating patterns and regular exercise for 12 weeks.

SUMMARY:
The aim of this study is To evaluate the impact of lifestyle modifications, including dietary changes and regular exercise, on skin-related quality of life in patients with pemphigus by assessing changes in Skindex-16 scores over a three-month period.

DETAILED DESCRIPTION:
The skin, the body's largest organ, serves as a critical protective barrier against environmental hazards and plays a pivotal role in immune defence.

Autoimmune diseases arise when the immune system erroneously targets the body's own tissues, leading to chronic inflammation and tissue damage. Globally, the prevalence of these disorders is on the rise, significantly impacting patient morbidity and healthcare systems.

Pemphigus is a rare autoimmune blistering disorder characterized by the production of autoantibodies against desmogleins-proteins essential for cell-to-cell adhesion within the epidermis.

Epidemiologically, pemphigus vulgaris (PV) is the most common subtype, with incidence rates varying geographically. Higher incidences are observed in regions such as the Middle East, with Iran reporting up to 5 cases per 100,000 people annually. In the Arab world, PV predominates in countries like Egypt, Sudan, and Morocco.

Complications of pemphigus are multifaceted. Patients are susceptible to secondary bacterial, viral, and fungal infections due to compromised skin integrity, which can escalate to sepsis. Oral mucosal involvement often leads to painful erosions, causing difficulties in alimentation and subsequent nutritional deficiencies.

The psychological burden of pemphigus is considerable. Chronic pain, visible lesions, and social stigma contribute to elevated rates of anxiety and depression among patients. Studies indicate that approximately 30.7% of individuals with pemphigus experience anxiety or depressive disorders, underscoring the need for comprehensive psychosocial support in this population.

Therapeutically, systemic corticosteroids remain the cornerstone of pemphigus management, often supplemented with immunosuppressants and biologic agents like rituximab. While effective, these treatments carry risks; long-term corticosteroid use is associated with adverse effects such as osteoporosis, increased infection risk, and metabolic disturbances.

Despite advancements in therapeutic strategies, there remains a paucity of research focusing on lifestyle modifications as adjunctive measures in managing pemphigus. This study aims to explore the potential benefits of integrating lifestyle interventions to enhance patient outcomes, reduce treatment-related complications, and improve overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18-65 years diagnosed with pemphigus. 2. Willingness and ability to adhere to prescribed lifestyle modifications.

Exclusion Criteria:

* 1. Presence of severe comorbidities that could impede adherence to dietary interventions and regular exercise 2. Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation the impact of lifestyle modifications, including dietary changes and regular exercise, on skin-related quality of life in patients with pemphigus by assessing changes in Skindex-16 scores over a three-month period | over a three-month period

SECONDARY OUTCOMES:
Prevalence of pemphigus in Assuit city | over 2 years